CLINICAL TRIAL: NCT01327885
Title: A Randomized, Open-label, Multicenter, Phase 3 Study to Compare the Efficacy and Safety of Eribulin With Dacarbazine in Subjects With Soft Tissue Sarcoma
Brief Title: Phase 3 Study to Compare the Efficacy and Safety of Eribulin With Dacarbazine in Subjects With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-309; 2010-024483-17 (EudraCT Number)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2018-02

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Eribulin mesylate 1.4 mg/m^2 intravenous
- Arm B (Active Comparator)
  Interventions: Drug: Dacarbazine of 850 mg/m^2, or 1,000 mg/m^2, or 1,200 mg/m^2 IV

INTERVENTIONS:
Drug: Eribulin mesylate 1.4 mg/m^2 intravenous — Administration of eribulin mesylate at a dose of 1.4 mg/m^2 as an intravenous (IV) bolus infusion over 2-5 minutes on Days 1 and 8 of every cycle, where the duration of each cycle is 21 days.
  Arms: Arm A
Drug: Dacarbazine of 850 mg/m^2, or 1,000 mg/m^2, or 1,200 mg/m^2 IV — Administration of dacarbazine at a dose of 850 mg/m^2, or 1,000 mg/m^2, or 1,200 mg/m^2 selected by the Principal Investigator [PI] or designee according to the subject's clinical status as an IV infusion over 15-30 minutes on Day 1 of every cycle, where the duration of each cycle is 21 days.
  Arms: Arm B

SUMMARY:
This is a randomized, open-label, multicenter, Phase 3 study comparing the efficacy and safety of eribulin with dacarbazine in subjects with advanced soft tissue sarcoma who have disease progression within 6 months prior to study enrolment following standard therapies which must have included an anthracycline, unless contraindicated and then at least one additional regimen after failure of the anthracycline.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of soft tissue sarcoma of high or intermediate grade with one of the following histological subtypes:

   * Adipocytic sarcoma, including:
   * Dedifferentiated
   * Myxoid
   * Round Cell
   * Pleomorphic - Leiomyosarcoma
2. Documented evidence of advanced (locally recurrent, locally advanced and/or metastatic) adipocytic (restricted to subtypes listed in Inclusion 1) or leiomyosarcoma, incurable by surgery and/or radiotherapy.
3. Subjects should have received at least two standard systematic regimens for advanced soft tissue sarcoma one of which must have included an anthracycline (unless contraindicated).
4. Radiographic evidence of disease progression by RECIST criteria on or after the last anti-cancer therapy within the 6 months prior to randomization.
5. Presence of measurable disease meeting the following criteria:

   * At least one lesion of greater than or equal to 1.0 cm in long-axis diameter for non lymph nodes or greater than or equal to 1.5 cm in short-axis diameter for lymph nodes which is serially measurable according to RECIST 1.1 using either computerized tomography or magnetic resonance imaging or panoramic and close-up color photography.
   * Lesions that have had radiotherapy must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
6. Eastern Cooperative Oncology Group, performance status of 0, 1 or 2.
7. Adequate renal function defined as calculated creatinine clearance greater than 50 mL/min per the Cockroft and Gault formula.
8. Adequate bone marrow function, defined as:

   * Absolute neutrophil count (ANC) greater than or equal to 1,500/mm3 or greater than or equal to 1.5 x 10^9/L.
   * Platelet count greater than or equal to 100,000/mm3 or greater than or equal to 100 x 10^9/L.
   * Hemoglobin (Hb) greater than or equal to 10g/dL at baseline (blood transfusions,hematopoietic growth factors and hematinics are allowed during the Prerandomization Phase to correct Hb values less than 10g/dL).
9. Adequate liver function, defined as:

   * Bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome.
   * Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times ULN. For total ALP greater than 3 times ULN, the ALP liver isoenzyme must be less than or equal to 3 times ULN.
10. All female subjects will be considered to be of child-bearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically (i.e., bilateral tubal ligation greater than or equal to 1 menstrual cycle prior to randomization, or have undergone a hysterectomy and/or bilateral oophorectomy).

    Female subjects of child-bearing potential must agree to use two forms of highly effective contraception from the last menstrual period prior to randomization (or use a double barrier method as described below until they are on two forms of highly effective contraception for at least one menstrual cycle), during the study treatment, and for 3 months after the final dose of study treatment. Female subjects exempt from this requirement are subjects who practice total abstinence. If currently abstinent, the subject must agree to use a double barrier method of contraception, i.e., condom and occlusive cap (diaphragm or cervical/vault caps) with spermicide or until they are on two forms of highly effective contraception for at least one menstrual cycle if they become sexually active during the study treatment and for 3 months after the final dose of study treatment. Highly effective contraception includes:
    * Placement of intrauterine device or system,
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) with spermicide,
    * Established hormonal contraceptive methods: oral, injectable or implant. Female subjects who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product from the last menstrual period prior to randomization, and must continue to use the same hormonal contraceptive product during study treatment, and for 3 months after the first dose of study treatment.
    * Vasectomized partner with confirmed azoospermia.
11. Male subjects and their female partner who are of child-bearing potential (as defined in Inclusion 10), and are not practicing total abstinence, must agree to use two forms of highly effective contraception from the last menstrual period of their female partner prior to randomization (or use a double barrier method as described above until they are on two forms of highly effective contraception for at least one menstrual cycle), during study treatment, and for 3 months (or 6 months if they received dacarbazine) after the final dose of study treatment. If currently abstinent, must agree to use a double barrier method of contraception if they become sexually active, or until they are on two forms of highly effective contraception as described above.
12. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.
13. Males or females aged greater than or equal to 18 years at the time of informed consent.

Exclusion Criteria:

1. Subjects who have received any anti-cancer therapy, including radiotherapy, cytotoxic, hormonal, biological (including humanized antibodies) and targeted agents within 21 days, or five half-lives of the drug (whichever is longer) prior to randomization.
2. Subjects who have not recovered from acute toxicities as a result of prior anti-cancer therapy to less than or equal to Grade 1, according to Common Terminology Criteria for Adverse Events (CTCAE), except for peripheral neuropathy (see Exclusion 6) and alopecia.
3. Subjects that have previously been treated with dacarbazine or its analogue temozolomide or eribulin.
4. Major surgery within 21 days prior to randomization.
5. Pre-existing peripheral neuropathy greater than CTCAE Grade 2.
6. Significant cardiovascular impairment, defined as:

   * Cardiac failure, New York Heart Association (NYHA) Class II according to the NYHA Functional Classification,
   * Unstable angina or myocardial infarction within 6 months of enrolment,
   * Serious and potentially life-threatening arrhythmia.
7. Subjects with a high probability of Long QT Syndrome or QTc interval prolongation of more than or equal to 501 msec on at least two separate ECGs, following correction of any electrolyte imbalance.
8. Subjects with known central nervous system metastases.
9. Any serious concomitant illness or infectious disease requiring treatment, or infectious disease not requiring treatment, but with significant risks for myelosuppressive complications associated with chemotherapy.
10. Any malignancy that required treatment, or has shown evidence of recurrence (except for soft tissue sarcoma, non-melanoma skin cancer, or histologically confirmed complete excision of carcinoma in situ) during the 5 years prior to randomization.
11. Female subjects must not be pregnant as documented by a negative beta-human chorionic gonadotropin (beta-hCG) test with a minimum sensitivity 25 IU/L or equivalent unit of beta-hCG at Screening and Baseline, or breastfeeding.
12. Hypersensitivity to the active substance, or any of the excipients of the eribulin drug product, or dacarbazine, (please refer to the dacarbazine prescribing information).
13. Any medical or other condition which, in the opinion of the PI or designee, will preclude participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2015-01-02 (Actual); Study Completion 2016-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (119):
- United States (30):
  - Tucson, Arizona
  - Los Angeles, California
  - Orange, California
  - Santa Monica, California
  - Stanford, California
  - Aurora, Colorado
  - Denver, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Atlanta, Georgia
  - Post Falls, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Urbana, Illinois
  - Iowa City, Iowa
  - Boston, Massachusetts
  - St Louis, Missouri
  - Newark, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Burlington, Vermont
  - Seattle, Washington
- Argentina (3):
  - Ciudad de Buenos Aires
  - San Miguel de Tucumán
  - San Salvador de Jujuy
- Australia (5):
  - Camperdown, New South Wales
  - St Leonards, New South Wales
  - Woolloongabba, Queensland
  - Woodville South, South Australia
  - Nedlands, Western Australia
- Austria (3):
  - Graz
  - Salzburg
  - Vienna
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Brazil (8):
  - Porto Alegre, Rio Grande do Sul
  - Florianópolis, Santa Catarina
  - Barretos
  - Curitiba
  - Jaú
  - Porto Alegre
  - Salvador
  - São Paulo
- Canada (3):
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (4):
  - Brno
  - Hradec Králové
  - Nový Jičín
  - Prague
- Herlev, Denmark
- France (9):
  - Angers
  - Bordeaux
  - Lyon
  - Marseille
  - Nantes
  - Paris
  - Poitiers
  - Saint-Priest-en-Jarez
  - Villejuif
- Germany (7):
  - Berlin
  - Cologne
  - Dresden
  - Essen
  - Hanover
  - Mannheim
  - Tübingen
- Israel (4):
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Italy (7):
  - Aviano, Pordenone
  - Candiolo
  - Milan
  - Monza
  - Padua
  - Rozzano (MI)
  - Torino
- Netherlands (2):
  - Amsterdam
  - Leiden
- Christchurch, New Zealand
- Poland (3):
  - Gdansk
  - Gliwice
  - Warsaw
- Romania (4):
  - Cluj-Napoca
  - Craiova
  - Iași
  - Sibiu
- Russia (4):
  - Chelyabinsk
  - Kazan'
  - Moscow
  - Obninsk
- Singapore, Singapore
- South Korea (3):
  - Daejeon
  - Seongnam
  - Seoul
- Spain (6):
  - Palma de Mallorca, Balearic Islands
  - Badalona, Catalonia
  - L'Hospitalet de Llobregat, Catalonia
  - Madrid, Madrid
  - Barcelona
  - Valencia
- Thailand (4):
  - Hat Yai, Changwat Songkhla
  - Bangkok
  - Chiang Mai
  - Pathum Wan
- United Kingdom (4):
  - Glasgow
  - London
  - Manchester
  - Swansea

REFERENCES:
- [Derived] Schoffski P, Chawla S, Maki RG, Italiano A, Gelderblom H, Choy E, Grignani G, Camargo V, Bauer S, Rha SY, Blay JY, Hohenberger P, D'Adamo D, Guo M, Chmielowski B, Le Cesne A, Demetri GD, Patel SR. Eribulin versus dacarbazine in previously treated patients with advanced liposarcoma or leiomyosarcoma: a randomised, open-label, multicentre, phase 3 trial. Lancet. 2016 Apr 16;387(10028):1629-37. doi: 10.1016/S0140-6736(15)01283-0. Epub 2016 Feb 10. PMID 26874885

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Eribulin Mesylate: Eribulin mesylate at a dose of 1.4 milligram per square meter (mg/m^2) was administered intravenously (IV) as a bolus infusion over 2-5 minutes on Days 1 and 8 of every 21-day treatment cycle.
- Arm B: Dacarbazine: Dacarbazine at a dose of 850 mg/m^2, 1000 mg/m^2, or 1200 mg/m^2 (as selected by the Principal Investigator [PI] or designee prior to randomization according to the participant's clinical status) was administered as an IV infusion over 15-30 minutes (or up to 60 minutes as per institutional guidelines) on Day 1 of every 21-day treatment cycle.
Period: Overall Study
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine
Started | 228 | 224
Completed | 0 | 0
Not Completed | 228 | 224
Not completed — Disease progression-according to RECIST | 173 | 165
Not completed — Clinical progression | 24 | 27
Not completed — Adverse Event | 14 | 10
Not completed — Subject choice | 5 | 10
Not completed — Other | 8 | 6
Not completed — Withdrawal of consent from study | 3 | 4
Not completed — Not treated | 1 | 1
Not completed — Administrative decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) (Intent-to-Treat (ITT) analysis set) included all participants who were randomized.
Groups:
- Arm A: Eribulin Mesylate: Eribulin mesylate at a dose of 1.4 mg/m^2 was administered IV as a bolus infusion over 2-5 minutes on Days 1 and 8 of every 21-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine | Total
Number analyzed (Participants) | 228 | 224 | 452
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 55.6 (11.01) | 55.7 (10.35) | 55.7 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 142 | 303
  Male | 67 | 82 | 149

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time in months from the date of treatment start until death, regardless of cause. In the absence of confirmation of death, participants were censored either at the date that participant was last known to be alive or the date of study cut-off, whichever was earlier. Participants who died on the date of randomization had a survival time of 0.5 day. Allocation of randomization numbers were performed based upon the following stratification factors: (a) Histology (adipocytic [ADI] or leiomyosarcoma [LMS]), (b) Region (Region 1: USA and Canada; or Region 2: Western Europe, Australia, Israel; or Region 3: Eastern Europe, Latin America, and Asia), and (c) Number of prior regimens for advanced soft tissue sarcoma (STS) (2 or greater than [>] 2 prior regimens).
Time Frame: From date of treatment start until date of death from any cause, up to 5 years 5 months
Population: Full analysis set (FAS) (Intent-to-Treat (ITT) analysis set) included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine
Number analyzed (Participants) | 228 | 224
Months | 13.5 [10.9 to 15.6] | 11.5 [9.6 to 13.0]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Dacarbazine; Statistical analysis was designed to detect superiority of Arm A (eribulin) over Arm B (dacarbazine). OS was compared between the two treatment arms using a two-sided stratified log-rank test at a nominal significance level of 0.0455 (adjusted for the interim analysis). This was the primary analysis that was performed when the target number of events (~353 deaths) was observed; Test type: Superiority or Other; p = 0.0169, Log Rank — The P-value was calculated by 2-sided log-rank test as stratified by histology, geographic region, and number of prior regimens for advanced STS; Hazard Ratio (HR) = 0.768, 95% CI 2-sided [0.618 to 0.954] — The Hazard Ratio is based on a stratified Cox regression model including treatment as covariate, and histology, geographic region, and number of prior regimens for advanced STS as strata

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of disease progression, or date of death (whichever occurred first). The date of disease progression was defined as the date of radiologic disease progression as assessed by the investigator or designee based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Participants who did not have an event (i.e., participants who were lost to follow-up or who did not progress or die at the date of data cut-off), were censored. Participants who discontinued study treatment without disease progression were censored on the date of their last radiological assessment (scan date).
Time Frame: Randomization (day 1) to the date of first documentation of disease progression, or date of death (whichever occurred first), up to 5 years 5 months
Population: FAS (ITT analysis set) included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm B: Dacarbazine: Dacarbazine at a dose of 850 mg/m^2, 1000 mg/m^2, or 1200 mg/m^2 (as selected by the PI or designee prior to randomization according to the participant's clinical status) was administered as an IV infusion over 15-30 minutes (or up to 60 minutes as per institutional guidelines) on Day 1 of every 21-day treatment cycle.
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine
Number analyzed (Participants) | 228 | 224
Months | 2.6 [1.9 to 2.8] | 2.6 [1.8 to 2.7]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Dacarbazine; The PFS and PFS rate at 3, 6, and 12 months (95% confidence interval (CI)) was calculated using Kaplan-Meier (K-M) product-limit method and Greenwood Formula. PFS was compared between the treatment arms using two-sided stratified log-rank test, stratified by histology, geographic region, and number of prior regimens for advanced STS; Test type: Superiority or Other; p = 0.2287, Log Rank — P-value was calculated by 2-sided log-rank test, as stratified by histology, geographic region, and number of prior regimens for advanced STS; Hazard Ratio (HR) = 0.877, 95% CI 2-sided [0.710 to 1.085] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Progression-Free Rate at 12 Weeks (PFR12wks)
Description: The PFR12wks was defined as the percentage of participants who were still alive without disease progression at 12 weeks from the date of randomization. Tumor assessment by the investigator or designee was based on RECIST criteria 1.1.
Time Frame: From date of randomization start until Week 12
Population: FAS (ITT analysis set) included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine
Number analyzed (Participants) | 228 | 224
Percentage of participants | 33.3 [27.2 to 39.9] | 28.6 [22.8 to 35.0]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Dacarbazine; The PFR12wks was compared between the treatment arms using stratified Cochran-Mantel-Haenszel (CMH) chi-square test stratified by histology, geographic region, and number of prior regimens for advanced STS; Test type: Superiority or Other; p = 0.253, Cochran-Mantel-Haenszel — The P-value was calculated using the stratified CMH method, the stratified factors included histology, geographic region, and number of prior regimens for advanced STS; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.8 to 1.9] — The odds ratio between eribulin and dacarbazine was calculated by stratified CMH method. The stratified factors were as described above. The 2-sided 95% CI of the odds ratio is based on asymptotic normal approximation

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants who have best overall response (BOR) of complete response (CR), or partial response (PR), or duration of stable disease (dSD) greater than or equal to 11 weeks, between Arm A and Arm B. CBR was estimated by treatment arm based on the tumor response evaluation performed by the PI or designee according to RECIST 1.1. CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter.
Time Frame: From date of treatment start (Day 1) until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice to stop study treatment, up to 5 years 5 months
Population: FAS (ITT analysis set) included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine
Number analyzed (Participants) | 228 | 224
Percentage of participants | 46.1 [39.5 to 52.8] | 47.8 [41.1 to 54.5]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Dacarbazine; The PFR12wks was compared between the treatment arms using stratified CMH chi-square test stratified by histology, geographic region, and number of prior regimens for advanced STS; Test type: Superiority or Other; p = 0.741, Cochran-Mantel-Haenszel — The P-value was calculated using the CMH method. The stratified factors were histology, geographic region, and number of prior regimens for advanced STS; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.7 to 1.4] — The Odds Ratio between eribulin and dacarbazine was calculated by stratified CMH method. The stratified factors were as described above. The 2-sided 95% CI of Odds Ratio is based on asymptotic normal approximation

ADVERSE EVENTS:
Time Frame: From date of signing of informed consent up to 30 days after the last dose of study treatment, up to 5 years 5 months
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Dacarbazine
All-Cause Mortality (participants affected / at risk) | 198/228 | 206/224
Serious Adverse Events (participants affected / at risk) | 76/228 | 71/224
Other Adverse Events (participants affected / at risk) | 224/228 | 218/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Eribulin Mesylate (N=228) | Arm B: Dacarbazine (N=224)
Neutropenia (Blood and lymphatic system disorders) | 11 | 10
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Leukopenia (Blood and lymphatic system disorders) | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 13
Atrial fibrillation (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Intestinal obstruction (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 10 | 4
Asthenia (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 2 | 1
Fatigue (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 3 | 2
Lung infection (Infections and infestations) | 2 | 0
Peritonitis bacterial (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Serratia bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Eribulin Mesylate (N=228) | Arm B: Dacarbazine (N=224)
Neutropenia (Blood and lymphatic system disorders) | 95 | 51
Anaemia (Blood and lymphatic system disorders) | 66 | 68
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 60
Leukopenia (Blood and lymphatic system disorders) | 36 | 22
Lacrimation increased (Eye disorders) | 18 | 1
Nausea (Gastrointestinal disorders) | 91 | 106
Constipation (Gastrointestinal disorders) | 70 | 58
Abdominal pain (Gastrointestinal disorders) | 42 | 32
Vomiting (Gastrointestinal disorders) | 43 | 50
Diarrhoea (Gastrointestinal disorders) | 38 | 35
Stomatitis (Gastrointestinal disorders) | 31 | 11
Abdominal pain upper (Gastrointestinal disorders) | 19 | 13
Dyspepsia (Gastrointestinal disorders) | 18 | 7
Abdominal distension (Gastrointestinal disorders) | 16 | 12
Dry mouth (Gastrointestinal disorders) | 12 | 4
Fatigue (General disorders) | 98 | 86
Pyrexia (General disorders) | 58 | 28
Asthenia (General disorders) | 46 | 51
Oedema peripheral (General disorders) | 27 | 17
Urinary tract infection (Infections and infestations) | 23 | 11
Upper respiratory tract infection (Infections and infestations) | 20 | 9
Aspartate aminotransferase increased (Investigations) | 21 | 5
Neutrophil count decreased (Investigations) | 19 | 12
Alanine aminotransferase increased (Investigations) | 18 | 8
White blood cell count decreased (Investigations) | 16 | 15
Electrocardiogram QT prolonged (Investigations) | 14 | 11
Blood lactate dehydrogenase increased (Investigations) | 12 | 7
Platelet count decreased (Investigations) | 2 | 17
Decreased appetite (Metabolism and nutrition disorders) | 43 | 43
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 46 | 8
Headache (Nervous system disorders) | 41 | 21
Dizziness (Nervous system disorders) | 21 | 16
Paraesthesia (Nervous system disorders) | 20 | 7
Dysgeusia (Nervous system disorders) | 18 | 5
Insomnia (Psychiatric disorders) | 22 | 10
Anxiety (Psychiatric disorders) | 12 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 33
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 79 | 6
Hypotension (Vascular disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No